CLINICAL TRIAL: NCT03153293
Title: A Single Intravitreal Injection of rAAV2-ND4 for the Treatment of Leber's Hereditary Optic Neuropathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Taihe Hospital (Other)
Responsible Party: Principal Investigator, Bin Li, professor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Leber 2
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Leber Hereditary Optic Neuropathy
Keywords: LHON,G11778A mutation, rAAV2-ND4，gene therapy
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rAAV2-ND4 (Experimental): A Single IVT Injection of recombinant Adeno-Associated Virus-NADH dehydrogenase, subunit 4 (complex I)（rAAV2-ND4)（0.05ml).The dose is 1 × 10^10 vg/0.05 mL for test groups.
  Interventions: Drug: rAAV2-ND4

INTERVENTIONS:
Drug: rAAV2-ND4 — a Single IVT Injection

SUMMARY:
This study is meant to evaluate the safety and efficacy of rAAV2-ND4 treatment for Leber hereditary optic neuropathy with the G11778A mutation in mitochondrial DNA.

DETAILED DESCRIPTION:
Leber's Optic Hereditary Neuropathy (LHON) is a maternally inherited ocular disorder primarily associated with mutations in mitochondrial DNA. The disease is a common cause of blindness in both eyes of affected teenagers and young adults. There is currently no approved effective treatment for LHON.

In 2011, the first LHON gene therapy investigator-initiated study was conducted (registered in December 2010 with ClinicalTrials.gov Identifier NCT01267422) to explore the safety and efficacy of gene therapy for LHON. The gene therapy was a recombinant adeno-associated virus serotype 2 containing human mitochondrial ND4 (MT-ND4) gene (rAAV2-ND4). By 36 months of follow-up, six out of nine patients who received the rAAV2-ND4 intravitreal injection experienced clinically significant vision improvement and no adverse events were observed.

This is an open-label, single-arm, multi-center study to further evaluate the safety and efficacy of rAAV-ND4 in the treatment of LHON patients with G11778A mutation. All patients will be treated with a single intravitreal injection rAAV-ND4, with dose 1 × 10^10 vg/0.05 mL in one of the eyes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients carry the mitochondrial point mutation at 11778, which is consistent with the diagnostic criteria for LHON.
2. No apparent eye sight improvement in LHON patients or any other treatment within the past year.
3. Eyesight of both eyes is below 0.3.
4. Patients signed written informed consent.
5. Patients are between the ages of 10 and 65 years old and able to tolerate the gene therapy procedure which includes local anesthesia.
6. Patients are willing to follow the doctor's instructions and to consult the doctor at prescribed times.
7. Patient's physical examination results are all normal, including liver function, kidney function, routine blood test, routine urine test, complete immunological test, and humoral immune response.

Exclusion Criteria:

1. Patients who are wearing a cardiac pacemaker, suffering from severe heart, lung or kidney function failure, various hemorrhagic diseases, acute infectious diseases, high fever, or convalescing after heart surgery or who are pregnant are excluded.
2. Patients who are participating in other clinical studies are excluded.
3. Patients who suffer from a diagnosed mental problem are excluded.
4. Patients who suffer from chronic diseases such as diabetes and hypertension are excluded.
5. Patients who show abnormal test results such as positive AAV2 humoral immune response (positive means that the AAV2 neutralizing antibody assay of patient was significant different when comparing free serum with 1:20 serum concentrations) and abnormal human T lymphocyte subsets CD3+, CD3+/CD4+ and CD3+/CD8+ prior to gene therapy surgery are excluded.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
BCVA | Change from Baseline at 12 months .
  The Best Corrected Visual Acuity
Computerized Visual Field | Change from Baseline at 12 months .

SECONDARY OUTCOMES:
VEP | Change from Baseline at 12 months .
  visual evoked potential
RNFL | Change from Baseline at 12 months .
  retinal nerve fiber layer
Liver function in plasma | Change from Baseline at 12 months .
kidney function in plasma | Change from Baseline at 12 months .

CONTACTS AND LOCATIONS:
Overall Officials: Bin Li, PhD,MD, Study Chair — Deputy Director of Ophthalmology,Tongji Hospital; Yong Zhang, PhD,MD, Principal Investigator — Director of Ophthalmology，Shiyan Taihe Hospital
Locations (1):
- Department of Ophthalmology，Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang S, Ma SQ, Wan X, He H, Pei H, Zhao MJ, Chen C, Wang DW, Dong XY, Yuan JJ, Li B. Long-term outcomes of gene therapy for the treatment of Leber's hereditary optic neuropathy. EBioMedicine. 2016 Aug;10:258-68. doi: 10.1016/j.ebiom.2016.07.002. Epub 2016 Jul 6. PMID 27426279
- [Result] Yang S, Yang H, Ma SQ, Wang SS, He H, Zhao MJ, Li B. Evaluation of Leber's hereditary optic neuropathy patients prior to a gene therapy clinical trial. Medicine (Baltimore). 2016 Oct;95(40):e5110. doi: 10.1097/MD.0000000000005110. PMID 27749593
- [Result] Ran R, Yang S, He H, Ma S, Chen Z, Li B. A retrospective analysis of characteristics of visual field damage in patients with Leber's hereditary optic neuropathy. Springerplus. 2016 Jun 23;5(1):843. doi: 10.1186/s40064-016-2540-7. eCollection 2016. PMID 27386292
- [Result] Wan X, Pei H, Zhao MJ, Yang S, Hu WK, He H, Ma SQ, Zhang G, Dong XY, Chen C, Wang DW, Li B. Efficacy and Safety of rAAV2-ND4 Treatment for Leber's Hereditary Optic Neuropathy. Sci Rep. 2016 Feb 19;6:21587. doi: 10.1038/srep21587. PMID 26892229
- [Result] Yang S, He H, Zhu Y, Wan X, Zhou LF, Wang J, Wang WF, Liu L, Li B. Chemical and material communication between the optic nerves in rats. Clin Exp Ophthalmol. 2015 Nov;43(8):742-8. doi: 10.1111/ceo.12547. Epub 2015 Jun 25. PMID 25950380
- [Result] Pei H, Wan X, Hu W, Dong X, Li B. Construction and detection of a novel type of recombinant human rAAV2/2-ND4. Eye Sci. 2013 Jun;28(2):55-9. PMID 24396955
- [Result] Cui G, Ding H, Xu Y, Li B, Wang DW. Applications of the method of high resolution melting analysis for diagnosis of Leber's disease and the three primary mutation spectrum of LHON in the Han Chinese population. Gene. 2013 Jan 1;512(1):108-12. doi: 10.1016/j.gene.2012.09.110. Epub 2012 Oct 9. PMID 23063736
- [Result] Shi H, Gao J, Pei H, Liu R, Hu WK, Wan X, Li T, Li B. Adeno-associated virus-mediated gene delivery of the human ND4 complex I subunit in rabbit eyes. Clin Exp Ophthalmol. 2012 Dec;40(9):888-94. doi: 10.1111/j.1442-9071.2012.02815.x. Epub 2012 Jul 2. PMID 22612072
- [Result] Feuer WJ, Schiffman JC, Davis JL, Porciatti V, Gonzalez P, Koilkonda RD, Yuan H, Lalwani A, Lam BL, Guy J. Gene Therapy for Leber Hereditary Optic Neuropathy: Initial Results. Ophthalmology. 2016 Mar;123(3):558-70. doi: 10.1016/j.ophtha.2015.10.025. Epub 2015 Nov 19. PMID 26606867
- [Result] Erickson RP. Leber's optic atrophy, a possible example of maternal inheritance. Am J Hum Genet. 1972 May;24(3):348-9. No abstract available. PMID 5063796
- [Result] Wallace DC, Singh G, Lott MT, Hodge JA, Schurr TG, Lezza AM, Elsas LJ 2nd, Nikoskelainen EK. Mitochondrial DNA mutation associated with Leber's hereditary optic neuropathy. Science. 1988 Dec 9;242(4884):1427-30. doi: 10.1126/science.3201231.
- [Result] Huoponen K, Vilkki J, Aula P, Nikoskelainen EK, Savontaus ML. A new mtDNA mutation associated with Leber hereditary optic neuroretinopathy. Am J Hum Genet. 1991 Jun;48(6):1147-53. PMID 1674640
- [Result] Mackey D, Howell N. A variant of Leber hereditary optic neuropathy characterized by recovery of vision and by an unusual mitochondrial genetic etiology. Am J Hum Genet. 1992 Dec;51(6):1218-28. PMID 1463007
- [Result] Maguire AM, Simonelli F, Pierce EA, Pugh EN Jr, Mingozzi F, Bennicelli J, Banfi S, Marshall KA, Testa F, Surace EM, Rossi S, Lyubarsky A, Arruda VR, Konkle B, Stone E, Sun J, Jacobs J, Dell'Osso L, Hertle R, Ma JX, Redmond TM, Zhu X, Hauck B, Zelenaia O, Shindler KS, Maguire MG, Wright JF, Volpe NJ, McDonnell JW, Auricchio A, High KA, Bennett J. Safety and efficacy of gene transfer for Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2240-8. doi: 10.1056/NEJMoa0802315. Epub 2008 Apr 27. PMID 18441370
- [Result] Bainbridge JW, Smith AJ, Barker SS, Robbie S, Henderson R, Balaggan K, Viswanathan A, Holder GE, Stockman A, Tyler N, Petersen-Jones S, Bhattacharya SS, Thrasher AJ, Fitzke FW, Carter BJ, Rubin GS, Moore AT, Ali RR. Effect of gene therapy on visual function in Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2231-9. doi: 10.1056/NEJMoa0802268. Epub 2008 Apr 27. PMID 18441371
- [Result] Hauswirth WW, Aleman TS, Kaushal S, Cideciyan AV, Schwartz SB, Wang L, Conlon TJ, Boye SL, Flotte TR, Byrne BJ, Jacobson SG. Treatment of leber congenital amaurosis due to RPE65 mutations by ocular subretinal injection of adeno-associated virus gene vector: short-term results of a phase I trial. Hum Gene Ther. 2008 Oct;19(10):979-90. doi: 10.1089/hum.2008.107. PMID 18774912
- [Result] Hufnagel RB, Ahmed ZM, Correa ZM, Sisk RA. Gene therapy for Leber congenital amaurosis: advances and future directions. Graefes Arch Clin Exp Ophthalmol. 2012 Aug;250(8):1117-28. doi: 10.1007/s00417-012-2028-2. Epub 2012 May 29. PMID 22644094
- [Result] Howell N, Bindoff LA, McCullough DA, Kubacka I, Poulton J, Mackey D, Taylor L, Turnbull DM. Leber hereditary optic neuropathy: identification of the same mitochondrial ND1 mutation in six pedigrees. Am J Hum Genet. 1991 Nov;49(5):939-50. PMID 1928099
- [Derived] Zhang Y, Yuan JJ, Liu HL, Tian Z, Liu SW, Li B. Three Cases of Leber's Hereditary Optic Neuropathy with Rapid Increase in Visual Acuity After Gene Therapy. Curr Gene Ther. 2019;19(2):134-138. doi: 10.2174/1566523219666190618094505. PMID 31237206